CLINICAL TRIAL: NCT03110172
Title: Short-term Efficacy of Antidepressant in Patients Underwent TKA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalian Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Zhu Bin, Principal Investigator，Graduate Student, Dalian Municipal Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I84412001
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis Of Knee
Keywords: Osteoarthritis; Depression; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Depression; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: All patients will be randomly divided into two groups. The control group is going to be given celecoxib 200mg/24h to 2 weeks after operation. On the basis of the above scheme, the The treatment group will receive duloxetine 60mg/24h to 8 weeks after operation.
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- KSS scale (Active Comparator): Knee Society Score with Duloxetine Hydrochloride
  Interventions: Drug: Duloxetine Hydrochloride
- HAMD-17 scale (Active Comparator): Hamilton Depression Score with Duloxetine Hydrochloride
  Interventions: Drug: Duloxetine Hydrochloride
- SF-36 scale (Active Comparator): Medical Outcomes Study Short Form-36 score with Duloxetine Hydrochloride
  Interventions: Drug: Duloxetine Hydrochloride
- WOMAC scale (Active Comparator): Western Ontario and McMaster Universities Index with Duloxetine Hydrochloride
  Interventions: Drug: Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride — The treatment group will receive duloxetine 60mg/24h to 8 weeks after operation
  Other Names: Cymbalta

SUMMARY:
By taking certain antidepressant in early postoperative period，which is supposed to improve the psychological status of patients with osteoarthritis, explore the effect of certain antidepressant on the recovery of the early stage after the operation of knee joint replacement.

DETAILED DESCRIPTION:
In this study, the investigators are going to investigate the efficacy of Duloxetine on pain, physical function, mental health and quality of life in patients underwent TKAs.

The control group is going to be given celecoxib 200mg/24h to 2 weeks after operation.On the basis of the above scheme, the treatment group is going to receiving duloxetine 60mg/24h to 8 weeks after operation.HAMD-17 scale, KSS scale, SF-36 scale and WOMAC scale will be used to evaluate the two groups before and after operation for 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. No extra articular malformations are diagnosed and accord with Kellgren-Lawrence criteria
2. Primary TKA surgery,Varus is smaller than 20°
3. Always there is no history of mental illness, no history of relevant medicine
4. Be able to read and understand Chinese, with good communication skills
5. Voluntary participation in this clinical study

Exclusion Criteria:

1. Previous history of mental and psychological illness
2. With severe diseases in respiratory system, circulatory system or digestive system
3. Allergic to duloxetine and celecoxib

Ages: 51 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pain score of participants with Duloxetine as assessed by Western Ontario and McMaster Universities Index after 4 weeks of treatment. | up to 6 months
  A face-to-face questionnaire will be conducted by two trained interviewers
Function score of participants with Duloxetine as assessed by Knee Society Score after 4 weeks of treatment. | up to 6 months
  A face-to-face questionnaire will be conducted by two trained interviewers

SECONDARY OUTCOMES:
Pain score of participants with Duloxetine as assessed by Western Ontario and McMaster Universities Index after 8 weeks of treatment. | up to 6 months
  A face-to-face questionnaire will be conducted by two trained interviewers
Function score of participants with Duloxetine as assessed by Knee Society Score after 8 weeks of treatment. | up to 6 months
  A face-to-face questionnaire will be conducted by two trained interviewers

CONTACTS AND LOCATIONS:
Overall Officials: QI Zhiming, MD, Study Director — Dalian Municipal Central Hospital
Locations (1):
- Dalian municipal central hospital, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes